CLINICAL TRIAL: NCT06205277
Title: Predictors of Residual Tumor at Second Transurethral Resection for pT1 Non-muscle Invasive Bladder Cancer
Acronym: START
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Francesco Claps, MD, University of Trieste
Other Study IDs: 113/21
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer; Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pT1 NMIBC who underwent second TURBt: Patients with pT1 NMIBC who underwent second TURBt after a macroscopically completede first TURBt within 6-8 weeks
  Interventions: Procedure: Second TURBt

INTERVENTIONS:
Procedure: Second TURBt — Second TURBt for pT1 NMIBC as per current EAU Guidelines.

SUMMARY:
The START study is a multicentre retrospective project. The aim is to identify clinico-pathological predictors of residual tumor at time of second transurethral resection of bladder tumor (re-TURBt) and to identify well-selected candidates for a risk-adapted strategy in which this procedure could be safely spared.

DETAILED DESCRIPTION:
Background

Transurethral resection of bladder tumor (TURBt) is the standard procedure for bladder cancer (BCa) diagnosis and represents, at the same time, the most important therapeutic moment for patients with non muscle-invasive bladder cancer (NMIBC). A second or re-staging TURBt (re-TURBt), performed within 2 - 6 weeks from the initial TURBt, is currently recommended in all patients harboring tumor invasion into the lamina propria (pT1). The importance of re-TURBT lies not only in the inadequacy of the initial resection but also in its ability in providing additional prognostic information essential for risk-stratification refining.

However, it should be underlined that re-TURBt is an invasive and morbid procedure that severely affects patients' quality of life as it has to be performed on a elderly subset of patients that is maybe still suffering from the consequences of the previous surgery. Moreover, re-TURBt represents a costly procedure and a non-negligible source of logistic difficulties since it has to be scheduled within 2 to 6 weeks from the previous resection, making waiting lists longer especially for non-high-volume centers.

For all these reasons, not all the published literature agrees on the value of re-TURBt. Recently many authors focused their attention to this debated topic, questioning whether the technique used for resection, the timing of the resection itself, or the presence of CIS or the presence of detrusor muscle in the first sampling could impact on the presence of residual disease at second TURBt.

As a cornerstone in the management of high-risk NMIBC patients, recently it was pointed out as re-TURBt could be safely spared in some cases in favor of immediate conservative or radical treatments as timing a crucial crossroad in BCa landscape.

Here, a multicentre cohort of 321 patients found that the presence of detrusor muscle at first TURBt specimen, the absence of concomitant CIS and the en-bloc resection technique were independent predictors of negative histology at re-TURBt.

Bearing this in mind, the aim of this multicentre study is to identify predictors of residual tumor at re-TURBt and to further explore their clinical applicability within a risk-adapted strategy to identify patients who can be safely spared from this procedure.

Hypothesis Residual disease at time of re-TURBt has distinct patterns of presentation.

Study Aims To define clinico-pathological predictors of residual tumor at time of re-TURBt. To identify well-selected candidates for a risk-adapted strategy in which this procedure could be safely spared.

Outcome Measures Primary Objectives: to explore the rate of influence and the impact on residual tumor at re-TURBt among: clinical and demographic variables, preoperatory systemic inflammatory markers, surgical determinants, and pathological features.

Secondary Objectives: to test the applicability and validity of such predictors into a nomogram to identify who could be safely spared from re-TURBt.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing second TURBt (re-TURBt) for pT1LG/HG NMIBC after a macroscopically completed first TURBt (in patients with multiple lesions only the index lesion pT1 conditioning the indication of re-TURBt will be considered). Therefore, presence of residual tumor or not at time of re-TURBt will be assessed at site of previous pT1.
2. patients able to provide written informed consent;
3. clinical-localized non-metastatic disease (cN0, cM0).

Exclusion Criteria:

1. patients with clinical non-localized BCa (cN+, cM+);
2. patients with incomplete resection at time of first TURBt according to surgeon: macroscopic evidence of residual tumor, too long resection requiring a second-look will be excluded from the current study;
3. patients with incomplete clinical or demographic or pathological data;
4. patients who were unable to provide written informed consent;
5. patients who underwent urgency or emergency procedures in life-threating scenario

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All pT1 NMIBC patients after a macroscopically completed first TURBt who underwent second TURBt within 6-8 weeks as per current EAU Guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patients with histologically confirmed evidence of residual tumor at second TURBt | 6 to 8 weeks
  Patients with histologically confirmed evidence of residual tumor at second TURBt defined as any pT BCa

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste - Azienda Ospedaliera Universitaria Giuliano Isontina, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No